CLINICAL TRIAL: NCT05805228
Title: The Effect of Sexual Counseling on the Sexual Lives of Couples During Pregnancy and Postpartum Period.
Brief Title: Sexual Life of Couples During Pregnancy and Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ceyda Esen, nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ceydaes
Record Dates: First submitted 2023-02-28; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Related; Postpartum Sexual Dysfunction; Sexual Dysfunction
Keywords: sexual counseling; pregnancy; postpartum; Information-motivation-behavioral model
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Sex Counseling

STUDY DESIGN:
Intervention Model Description: This study was conducted with experimental and control group design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The sexual counseling program was applied to the couples in the experimental group in 2 sessions. The "Sexual Counseling I" session which includes information about sexual life specific to the pregnancy period, was conducted at least one week later the pre-test, with face-to-face interview method in a private room in the pregnancy outpatient clinic. The "Sexual Counseling II" session, which contains information on sexual life specific to the postpartum period, was conducted online in the third trimester of pregnancy with the video interview method. Counseling sessions consisted of power point presentations (including figures and drawings) and counseling booklet. The counseling booklet prepared by the researcher in accordance with literature consisted of two parts; sexual life during pregnancy and postpartum sexual life. Each session lasted 45 minutes and additional time was allocated for answering the questions.
  Interventions: Other: Sexual Counseling
- Control Group (No Intervention): Only routine antenatal and postnatal care was given to the couples in the control group

INTERVENTIONS:
Other: Sexual Counseling — Pregnancy and postpartum period-specific sexual counseling was given to pregnant women and their spouses.
  Arms: Experimental Group

SUMMARY:
The aim of this clinical trials is to determine the effect of sexual counseling applied in line with a special counseling model on the sexual functions of couples during pregnancy and postpartum period in order to prevent sexual problems that may occur in the pregnant woman and her husband during pregnancy.

The main questions it aims to answer are:

1. Does sexual counseling to be conducted during pregnancy prevent the problems that may occur in women during pregnancy and postpartum period?
2. Does sexual counseling to be conducted during pregnancy prevent the problems that may occur in pregnant women's husband during pregnancy and postpartum period? Questionnaires evaluating the sexual lives of the participants were administered. Afterwards, sexual counseling was given to the pregnant woman and her husband in the first three months of pregnancy. After the counseling, the questionnaires were applied again in the later stages of pregnancy and in the postpartum period. In order to see whether sexual counseling affects sexual problems that may develop during pregnancy and postpartum period, the researchers compared the counseling couples with the pregnant women who did not receive counseling and their spouses.

DETAILED DESCRIPTION:
Before starting the research, the researcher participated in the Sex Therapy Education Certificate Program to better research and educate pregnant women and their spouses. After she completed the certificate program, necessary permissions were obtained from the related institution. Verbal and written consent was obtained from the couples who came to the outpatient clinic for routine pregnancy monitoring at ten-fourteen weeks of pregnancy. The couples were interviewed through face-to-face interview method by applying the information form and scales in an appropriate environment that allows for privacy. Couples who met the criteria after pre-evaluation were included in the study. The separation of the groups was made by the medical secretary of the outpatient clinic, who was unrelated to the study, using a pre-coded list according to the order of arrival of the couples. Participants were divided into two groups as experimental and control. An appointment was made for the couples in the experimental group for an interview at a time convenient for them and in a suitable environment in the hospital. In accordance with IMB Model stages, a counseling for sexual health of the couples was planned and provided. The couples in the experimental group were given routine prenatal and postnatal care with sexual counseling. Only routine antenatal and postnatal care was given to the couples in the control group . The scales were applied to both groups four times in total, and repeated measurements were made. The scales were applied to both groups 4 times in total, in the first, second, third trimesters of pregnancy and in the 3rd month postpartum, and repeated measurements were made. All the scales after the first measurement were obtained by filling in the forms of the couples online. The couples in the experimental group were called by phone between each measurement and a total of three online interviews were made.

Sexual Counseling Process The sexual counseling program was applied to the couples in the experimental group in two sessions. The "Sexual Counseling I" session which includes information about sexual life specific to the pregnancy period, was conducted at least one week later the pre-test, with face-to-face interview method in a private room in the pregnancy outpatient clinic. The "Sexual Counseling II" session, which contains information on sexual life specific to the postpartum period, was conducted online in the third trimester of pregnancy with the video interview method. Counseling sessions consisted of power point presentations (including figures and drawings) and counseling booklet. The counseling booklet prepared by the researcher in accordance with literature consisted of two parts; sexual life during pregnancy and postpartum sexual life. Each session lasted forty-five minutes and additional time was allocated for answering the questions. After the counseling, the counseling booklets were given to the couples online. In addition, they were given a contact number where they could contact the consultant and ask questions, and they were contacted during the study.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid pregnant women at 10-14 weeks of gestation and their spouses
* Pregnant women and their spouses with FSFI Scale score ≤26.55
* Couples with regular sex life

Exclusion Criteria:

* Having a high-risk pregnancy
* Being pregnant with infertility treatment
* The couples had a history of medical illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Change From Baseline In Sexual Function On The Pregnant Women's Female Sexual Function Index (FSFI) Score Averages at 8 Months | baseline, 12 week after baseline, 8 week after second measurement and 12 week after third measurement
  FSFI is a validated. This index has nineteen items about sexual functioning of the patients during the last one month. High scores signify positive assessments. Total score of the scale ranges between two and thirty-six points. The scale's cutoff point is 26.55 and getting a score of 26.55 is considered to have sexual dysfunction. Change= baseline (14th week of pregnancy)-12 week after first measurement (28th week of pregnancy)- 8 week after second measurement (36th of week of pregnancy)- 12 week after third measurement (3rd month after delivery)
Change From Baseline In Sexual function On The Men With a Pregnant Wife On The Arizona Sexual Experiences Scale (ASEX) Score Averages of at 8 Months | baseline, 12 week after baseline, 8 week after second measurement and 12 week after third measurement
  This scale is a validated. This scale was developed to reveal and evaluate sexual functions and disorders in sexual functions. In the scale, each of the sexual functions in the last week is questioned with a question. It has 5 sub-scales: sexual desire, erection, orgasm and satisfaction. Each of the questions is scored between 1-6 points. The total scale score varies between 5 points and 30 points. High scores signify a low degree of sexual function. Change= baseline (14th week of pregnancy)-12 week after first measurement (28th week of pregnancy)- 8 week after second measurement (36th of week of pregnancy)- 12 week after third measurement (3rd month after delivery)
Change From Baseline In Sexual Satisfaction On The Pregnant Women's The New Sexual Satisfaction Scale Score Averages at 8 Months | baseline, 12 week after baseline, 8 week after second measurement and 12 week after third measurement
  This scale is a validated. These are the results of evaluating the sexual satisfactions of pregnant women. There are 20 items in the scale that can be scored between 1 and 5. The lowest score that can be obtained from the scale is 20, and the highest score is 100. The total scoring of the scale is calculated by summing the items. As the total score of the scale increases, the sexual satisfaction of the individual also increases. Change= baseline (14th week of pregnancy)-12 week after first measurement (28th week of pregnancy)- 8 week after second measurement (36th of week of pregnancy)- 12 week after third measurement (3rd month after delivery)
Change From Baseline In Sexual Satisfaction On The Men With a Pregnant Wife The New Sexual Satisfaction Scale Score Averages at 8 Months | baseline, 12 week after baseline, 8 week after second measurement and 12 week after third measurement
  This scale is a validated. These are the results of evaluating the sexual satisfactions of pregnant women's husband. There are 20 items in the scale that can be scored between 1 and 5. The lowest score that can be obtained from the scale is 20, and the highest score is 100. The total scoring of the scale is calculated by summing the items. As the total score of the scale increases, the sexual satisfaction of the individual also increases. Change= baseline (14th week of pregnancy)-12 week after first measurement (28th week of pregnancy)- 8 week after second measurement (36th of week of pregnancy)- 12 week after third measurement (3rd month after delivery)

SECONDARY OUTCOMES:
Change From Baseline In Depression Symptom Levels On The Pregnant Women The Center for Epidemiological Studies-Depression Scale Score Averages at 8 Months | baseline, 12 week after baseline, 8 week after second measurement and 12 week after third measurement
  This scale is a validated. The scale evaluates depressive symptoms and other variables that affect it. There are 20 items in the scale, each scored between 0-3 points. The scale questions the past week. The total score of the scale varies between 0-60 points. A score of 16 and above suggests the presence of depression. Change= baseline (14th week of pregnancy)-12 week after first measurement (28th week of pregnancy)- 8 week after second measurement (36th of week of pregnancy)- 12 week after third measurement (3rd month after delivery)
Change From Baseline In Depression Symptom Levels On The Men With a Pregnant Wife The Center for Epidemiological Studies-Depression Scale Score Averages at 8 Months | baseline, 12 week after baseline, 8 week after second measurement and 12 week after third measurement
  This scale is a validated. The scale evaluates depressive symptoms and other variables that affect it. There are 20 items in the scale, each scored between 0-3 points. The scale questions the past week. The total score of the scale varies between 0-60 points. A score of 16 and above suggests the presence of depression. Change= baseline (14th week of pregnancy)-12 week after first measurement (28th week of pregnancy)- 8 week after second measurement (36th of week of pregnancy)- 12 week after third measurement (3rd month after delivery)

CONTACTS AND LOCATIONS:
Overall Officials: ceyda esen, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- istanbul university Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alidost F, Pakzad R, Dolatian M, Abdi F. Sexual dysfunction among women of reproductive age: A systematic review and meta-analysis. Int J Reprod Biomed. 2021 Jun 23;19(5):421-432. doi: 10.18502/ijrm.v19i5.9251. eCollection 2021 May. PMID 34278195
- [Background] Alidost, F., Dolatian, M., Shams, J., Nasiri, M., Reisabdollahi, H., Pakzad, M.,ve diğ., 2021(b), The Relationship Between The Wealth Index And Pregnancy-Related Anxiety In Each Trimester Of Pregnancy And Their Effect On Sexual Dysfunction, Bangladesh Journal of Medical Science, 20, 401-408.
- [Background] Alizadeh S, Riazi H, Majd HA, Ozgoli G. The effect of sexual health education on sexual activity, sexual quality of life, and sexual violence in pregnancy: a prospective randomized controlled trial. BMC Pregnancy Childbirth. 2021 Apr 26;21(1):334. doi: 10.1186/s12884-021-03803-8. PMID 33902468
- [Background] Allen L, Fountain L. Addressing sexuality and pregnancy in childbirth education classes. J Perinat Educ. 2007 Winter;16(1):32-6. doi: 10.1624/105812407X171076. PMID 18408809
- [Background] Allsop DB, Leavitt CE, Yorgason JB, Holmes EK. Variable Sexual Satisfaction in Pregnancy: A Latent Profile Analysis of Pregnant Wives and Their Husbands. J Sex Res. 2022 Feb;59(2):173-184. doi: 10.1080/00224499.2021.1970708. Epub 2021 Sep 14. PMID 34520286
- [Background] Aslan G, Aslan D, Kizilyar A, Ispahi C, Esen A. A prospective analysis of sexual functions during pregnancy. Int J Impot Res. 2005 Mar-Apr;17(2):154-7. doi: 10.1038/sj.ijir.3901288. PMID 15538394
- [Background] Bahadoran P, MohammadiMahdiabadzade M, Nasiri H, GholamiDehaghi A. The effect of face-to-face or group education during pregnancy on sexual function of couples in Isfahan. Iran J Nurs Midwifery Res. 2015 Sep-Oct;20(5):582-7. doi: 10.4103/1735-9066.164512. PMID 26457096
- [Background] Bahrami Z, Zarani F. Application of the Information-Motivation and Behavioral Skills (IMB) model in risky sexual behaviors amongst male students. J Infect Public Health. 2015 Mar-Apr;8(2):207-13. doi: 10.1016/j.jiph.2014.09.005. Epub 2014 Nov 22. PMID 25466597
- [Background] Bakir E, Cavusoglu H, Mengen E. Effects of the Information-Motivation-Behavioral Skills Model on Metabolic Control of Adolescents with Type 1 Diabetes in Turkey: Randomized Controlled Study. J Pediatr Nurs. 2021 May-Jun;58:e19-e27. doi: 10.1016/j.pedn.2020.11.019. Epub 2020 Dec 25. PMID 33371976
- [Background] Baksu B, Davas I, Agar E, Akyol A, Varolan A. The effect of mode of delivery on postpartum sexual functioning in primiparous women. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Apr;18(4):401-6. doi: 10.1007/s00192-006-0156-0. Epub 2006 Jul 27. PMID 16871432
- [Background] Behzadipour, S., Daneshpour, M., Damreihani, N., Aflatooni, L., 2021, Sexual satisfaction and intimacy during pregnancy and after childbirth, Sexologies, 30,2, e111-e117.
- [Background] Bokaie M, Gashiri MZ, Khoshbin A, Salimi H. The effectiveness of sexual health counseling based on cognitive-behavioral therapy on sexual satisfaction and inefficient sexual beliefs of primigravida women. J Educ Health Promot. 2022 Feb 26;11:67. doi: 10.4103/jehp.jehp_521_20. eCollection 2022. PMID 35372614
- [Background] Cai Y, Ye X, Shi R, Xu G, Shen L, Ren J, Huang H. Predictors of consistent condom use based on the Information-Motivation-Behavior Skill (IMB) model among senior high school students in three coastal cities in China. BMC Infect Dis. 2013 Jun 4;13:262. doi: 10.1186/1471-2334-13-262. PMID 23734860
- [Background] Cattani L, De Maeyer L, Verbakel JY, Bosteels J, Deprest J. Predictors for sexual dysfunction in the first year postpartum: A systematic review and meta-analysis. BJOG. 2022 Jun;129(7):1017-1028. doi: 10.1111/1471-0528.16934. Epub 2021 Oct 17. PMID 34536325
- [Background] Chapa HO, Fish JT, Hagar C, Wilson T. Prevalence of female sexual dysfunction among women attending college presenting for gynecological care at a university student health center. J Am Coll Health. 2020 Jan;68(1):52-60. doi: 10.1080/07448481.2018.1515751. Epub 2018 Nov 2. PMID 30388952
- [Background] Dancet EAF, D'Hooghe TM, Dreischor F, van Wely M, Laan ETM, Lambalk CB, Repping S, Custers IM. The 'Pleasure&Pregnancy' web-based interactive educational programme versus expectant management in the treatment of unexplained subfertility: protocol for a randomised controlled trial. BMJ Open. 2019 Jul 9;9(7):e025845. doi: 10.1136/bmjopen-2018-025845. PMID 31289062
- [Background] Dabiri F, Yabandeh AP, Shahi A, Kamjoo A, Teshnizi SH. The effect of mode of delivery on postpartum sexual functioning in primiparous women. Oman Med J. 2014 Jul;29(4):276-9. doi: 10.5001/omj.2014.72. PMID 25170409
- [Background] Dagli E, Kul Uctu A, Ozerdogan N. Sexual dysfunction in the postpartum period: Its relationship with postpartum depression and certain other factors. Perspect Psychiatr Care. 2021 Apr;57(2):604-609. doi: 10.1111/ppc.12583. Epub 2020 Jul 17. PMID 32677049
- [Background] Dawson SJ, Leonhardt ND, Impett EA, Rosen NO. Associations Between Postpartum Depressive Symptoms and Couples' Sexual Function and Sexual Distress Trajectories Across the Transition to Parenthood. Ann Behav Med. 2021 Aug 23;55(9):879-891. doi: 10.1093/abm/kaaa117. PMID 33449076
- [Background] Evcili F, Demirel G, Bekar M, Guler H. Effectiveness of postpartum sexual health education programme structured according to Levine's conservation model: An interventional study. Int J Nurs Pract. 2020 Jun;26(3):e12855. doi: 10.1111/ijn.12855. Epub 2020 Jun 8. PMID 32510741
- [Background] Ge J, Wang L, Peng X, Zhang C, Zhao S, Zhou M, Tang S, You H. Behaviour model integrated by protection motivation theory and information-motivation-behavioural skills model applying in pregnancy weight management (PrInMAMa): a study protocol for a randomised controlled trial in China. BMJ Open. 2022 Jan 12;12(1):e051275. doi: 10.1136/bmjopen-2021-051275. PMID 35022170
- [Background] Gregory A. Understanding female sexual dysfunction, its causes and treatments. Br J Nurs. 2021 Oct 14;30(18):S18-S29. doi: 10.12968/bjon.2021.30.18.S18. PMID 34645346
- [Background] Gutzeit O, Levy G, Lowenstein L. Postpartum Female Sexual Function: Risk Factors for Postpartum Sexual Dysfunction. Sex Med. 2020 Mar;8(1):8-13. doi: 10.1016/j.esxm.2019.10.005. Epub 2019 Dec 16. PMID 31837965
- [Background] Heidari M, Aminshokravi F, Zayeri F, Azin SA. Effect of Sexual Education on Sexual Function of Iranian Couples During Pregnancy: A Quasi Experimental Study. J Reprod Infertil. 2018 Jan-Mar;19(1):39-48. PMID 29850446
- [Background] Jacob L, Smith L, Butler L, Barnett Y, Grabovac I, McDermott D, Armstrong N, Yakkundi A, Tully MA. Challenges in the Practice of Sexual Medicine in the Time of COVID-19 in the United Kingdom. J Sex Med. 2020 Jul;17(7):1229-1236. doi: 10.1016/j.jsxm.2020.05.001. Epub 2020 May 14. PMID 32411271
- [Background] John SA, Walsh JL, Weinhardt LS. The Information-Motivation-Behavioral Skills Model Revisited: A Network-Perspective Structural Equation Model Within a Public Sexually Transmitted Infection Clinic Sample of Hazardous Alcohol Users. AIDS Behav. 2017 Apr;21(4):1208-1218. doi: 10.1007/s10461-016-1446-2. PMID 27260181
- [Result] Afshar M, Mohammad-Alizadeh-Charandabi S, Merghti-Khoei ES, Yavarikia P. The effect of sex education on the sexual function of women in the first half of pregnancy: a randomized controlled trial. J Caring Sci. 2012 Nov 22;1(4):173-81. doi: 10.5681/jcs.2012.025. eCollection 2012 Dec. PMID 25276693
- [Result] Barrett G, Pendry E, Peacock J, Victor C, Thakar R, Manyonda I. Women's sexual health after childbirth. BJOG. 2000 Feb;107(2):186-95. doi: 10.1111/j.1471-0528.2000.tb11689.x. PMID 10688502